CLINICAL TRIAL: NCT00713531
Title: Cohort Study of HIV-1 Incidence Among Clients of the Thai Red Cross AIDS Research Center, Bangkok, Thailand
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Jintanat Ananworanich, SEARCH Research Foundation
Other Study IDs: SEARCH 008/RV233
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections
Keywords: HIV-negative; male and female clients; ages 18-50 years; seeking HIV counseling; testing at TRCARC
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, CD4, HIV-RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess populations in Thailand at high risk for HIV-1 infection for potential efficacy trials of candidate HIV vaccines to include:

1. assess incidence of HIV-1 and volunteer retention
2. describe early viral load and CD4 counts
3. assess participant willingness to participate in HIV vaccine efficacy trials and other HIV prevention trials
4. describe volunteer risk behavior

DETAILED DESCRIPTION:
Prospective cohort study of HIV-negative participants who will receive voluntary counseling and testing (VCT) for HIV-antibody in conjunction with questionnaires on risk behavior, willingness to participate in HIV vaccine trials and other HIV prevention trials at 4 month intervals for a period of 1 year. This study will follow 1000 HIV-negative volunteers with an expected minimum of 15-20 incident HIV-infections based on a minimum incidence rate of 1.5/100 person-years. Weighted incidence estimates will be calculated with exact 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18-50 years
* Willing to provide location or contact information and allow contact
* Thai citizenship as identified by Thai National Identification card
* Ability and willingness to provide consent
* Availability for follow-up for the planned study duration

Exclusion Criteria:

* Persons who have a history of a medical or psychiatric disorder, that in the judgment of the investigator(s), would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent
* Persons who are known to be HIV-positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Population in Thailand who are seeking HIV counseling and testing at TRCARC
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
number of HIV-1 infections per 100 person-years | 5 years
Lost to follow-up on an annual basis (10% or better) | 5 years
Post-infection viral load and CD4 count | 5 years
Willingness to participate in HIV vaccine and prevention trials | 5 years
Risk behavior by questionnaire | 5 years

SECONDARY OUTCOMES:
HIV-1 prevalence | 5 years
HIV-1 genotype distribution | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nittay - Phanuphak, MD., Principal Investigator — The Thai Red Cross AIDS Research Centre, Bangkok, Thailand
Locations (1):
- The Thai Red Cross AIDS Research Centre, Bangkok, Bangkok, Thailand